CLINICAL TRIAL: NCT02464228
Title: An Open Label Phase II Study of Tipifarnib in Subjects With Relapsed or Refractory Peripheral T-Cell Lymphoma
Brief Title: Investigation of Tipifarnib in Treatment of Subjects With Peripheral T-Cell Lymphoma (PTCL) That Have Not Responded to Standard Therapy
Acronym: PTCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kura Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KO-TIP-002
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-04

CONDITIONS: Relapsed or Refractory Peripheral T-Cell Lymphoma
Keywords: PTCL-NOS; Lymphoma; AITL; Nodal T-follicular helper phenotype; ALCL; Hepatosplenic T-cell lymphoma; EATL; Extranodal (NK) T-cell lymphoma; Wild Type CXCL12 3' UTR
MeSH Terms: conditions — Recurrence; Lymphoma, T-Cell, Peripheral; Lymphoma; Lymphoma, Extranodal NK-T-Cell | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tipifarnib (Experimental): tipifarnib, oral
  Interventions: Drug: Tipifarnib

INTERVENTIONS:
Drug: Tipifarnib — oral
  Other Names: Zarnesta

SUMMARY:
Phase II study designed to investigate antitumor activity in terms of objective response rate (ORR) of tipifarnib subjects with advanced Peripheral T-Cell Lymphoma (PTCL). Tipifarnib will be administered orally until disease progression.

DETAILED DESCRIPTION:
This Phase II study will investigate the antitumor activity in terms of ORR of tipifarnib in subjects with relapsed or refractory PTCL. The first 18 subjects may be of the following PTCL sub-types: PTCL not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), ALK-positive and negative anaplastic large cell lymphoma (ALCL), hepatosplenic T-cell lymphoma, enteropathy-associate T-cell lymphoma (EATL), extranodal natural killer (NK) T-cell lymphoma, nasal type and subcutaneous panniculitis-like T-cell lymphoma. The AITL expansion cohort (N=32) will enroll only subjects with AITL. An additional cohort of patients (N=12) expressing the wild type CXCL12 3' UTR will be enrolled in order to explore the benefits of tipifarnib treatment observed in patients having an absence of this gene variation or single nucleotide variation (SNV).

Tumor response assessments will be conducted according to Lugano Classification and/or mSWAT criteria.

Tumor assessments will be performed approximately every 8 weeks (cycles 2-6) and at least once approximately every 12 weeks thereafter (Cycles 9, 12, 15, etc.), and will continue until disease progression. Subjects experiencing a complete response may be considered for bone marrow transplantation. Upon disease progression, all subjects will be followed for survival and the use of subsequent therapy. All subjects will be followed for safety during treatment and up to approximately 30 days after treatment discontinuation or until before the initiation of another anti-cancer therapy. Additional follow up may be implemented until the subject recovers from any emergent treatment related toxicity or the adverse event is considered irreversible by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PTCL according to the most recent edition of the World Health Organization (WHO) Classification of Tumors of Hematopoietic or Lymphoid Tissues, as follows:

   1. Anaplastic large cell lymphoma (ALCL), ALK positive
   2. ALCL, ALK negative
   3. Angioimmunoblastic T-cell lymphoma (AITL)
   4. Enteropathy-associated T-cell lymphoma
   5. Extranodal natural killer (NK) T-cell lymphoma, nasal type
   6. Hepatosplenic T-cell lymphoma
   7. Peripheral T-cell lymphoma, not otherwise specified (NOS)
   8. Subcutaneous panniculitis-like T-cell lymphoma
2. For enrollment into the AITL expansion cohort, subjects must have the diagnosis of AITL, nodal PTCL with T-follicular helper phenotype or follicular PTC.
3. For enrollment into the CXCL12+ PTCL expansion cohort, subjects must have the diagnosis of PTCL (a - h subtypes listed above, except AITL), consent to provide buccal swabs for CXCL12 SNP testing, and be found to be CXCL12+ based on testing by a Sponsor approved methodology.
4. Relapsed or are refractory to at least 1 prior systemic cytotoxic therapy. -Subjects must have received conventional therapy as a prior therapy.
5. Subject has consented to provide at least 6 unstained tumor slides (10 preferred) or an FFPE block for biomarker testing.
6. Subject has measurable disease as determined by the Lugano Classification and/or mSWAT.
7. At least 2 weeks since the last systemic therapy regimen prior to enrollment.
8. At least 2 weeks since last radiotherapy if radiation was localized to the only site of measurable disease, unless there is documentation of disease progression of the irradiated site. Subjects must have recovered from all acute toxicities from radiotherapy.
9. ECOG performance status of 0-2
10. Acceptable liver and renal function
11. Acceptable hematologic status
12. Female subjects must be either:

    1. Of non-child-bearing potential (surgically sterilized or at least 2 years post- menopausal); or
    2. If of child-bearing potential, subject must use an adequate method of contraception consisting of two-barrier method or one barrier method with a spermicide or intrauterine device. Both females and male subjects with female partners of child- bearing potential must agree to use an adequate method of contraception for 2 weeks prior to screening, during, and at least 4 weeks after last dose of trial medication. Female subjects must have a negative serum or urine pregnancy test within 72 hours prior to start of trial medication.
    3. Not breast feeding at any time during the study.
13. Written and voluntary informed consent.

Exclusion Criteria:

1. Diagnosis of any of the following:

   1. Precursor T-cell lymphoma or leukemia
   2. Adult T-cell lymphoma/leukemia (ATLL)
   3. T-cell prolymphocytic leukemia
   4. T-cell large granular lymphocytic leukemia
   5. Primary cutaneous type anaplastic large cell lymphoma
   6. Mycosis fungoide/Sezary syndrome
2. Ongoing treatment with an anticancer agent not contemplated in this protocol.
3. Prior treatment (at least 1 full treatment cycle) with an FTase inhibitor.
4. Any history of clinically relevant coronary artery disease or myocardial infarction within the last 3 years.
5. Known central nervous system lymphoma.
6. Stem cell transplant less than 3 months prior to enrolment.
7. Non-tolerable > Grade 2 neuropathy or evidence of unstable neurological symptoms within 4 weeks of Cycle 1 Day 1.
8. Major surgery, other than diagnostic surgery, within 2 weeks prior to Cycle 1 Day 1, without complete recovery.
9. Other active malignancy requiring therapy such as radiation, chemotherapy, or immunotherapy.
10. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.

    Known infection with HIV, or an active infection with hepatitis B or hepatitis C.
11. Subjects who have exhibited allergic reactions to tipifarnib, or structural compounds similar to tipifarnib or to its excipients. This includes hypersensitivity to imidazoles, such as clotrimazole, ketoconazole, miconazole and others in this drug class.
12. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.
13. The subject has legal incapacity or limited legal capacity.
14. Dementia or significantly altered mental status that would limit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
15. Unwillingness or inability to comply with the study protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - Stanford University Medical Center, Palo Alto, California
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
- Samsung Medical Center, Seoul, South Korea
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia de Girona, Girona
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario 12 Octubre de Madrid, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Witzig T, Sokol L, Kim WS, de la Cruz Vicente F, Martin Garcia-Sancho A, Advani R, Roncero Vidal JM, de Ona Navarrete R, Marin-Niebla A, Rodriguez Izquierdo A, Terol MJ, Domingo-Domenech E, Saunders A, Bendris N, Mackey J, Leoni M, Foss F. Phase 2 trial of the farnesyltransferase inhibitor tipifarnib for relapsed/refractory peripheral T-cell lymphoma. Blood Adv. 2024 Sep 10;8(17):4581-4592. doi: 10.1182/bloodadvances.2024012806. PMID 38991123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 25 Feb 2016 (13 in Europe; 52 outside Europe) and the date of the last visit was 31 Mar 2021. Overall, 65 subjects were enrolled into cohorts with angioimmunoblastic T-cell lymphoma (AITL), peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS), PTCL-NOS whose tumors expressed high levels of C-X-C motif chemokine 12 (CXCL12+), and Other (anaplastic large cell lymphoma-anaplastic lymphoma kinase [ALCL-ALK negative] and PTCL-subtype not specified).
Pre-assignment Details: Only consented subjects who met all the eligibility criteria were enrolled in the study. All screening evaluations were to be completed within 4 weeks (28 days) of Cycle 1 Day 1. Screen failure reasons were not included in the database.
Groups:
- Cohort AITL: Subjects with AITL received tipifarnib as monotherapy. Tipifarnib was administered with food at a starting dose of 300 mg orally twice daily (BID) on Days 1 - 21 of 28-day treatment cycles.
  In the absence of unmanageable toxicity, treatment may have been continued as long as the investigator considered that the treatment was providing clinical benefit for up to 12 months since the subject's enrollment. Treatment may have continued beyond 12 months upon agreement by the investigator and sponsor if there was documented evidence of sustained clinical benefit.
- Cohort PTCL-NOS: Subjects with PTCL-NOS (not including subjects with PTCL-NOS CXCL12+) received tipifarnib as monotherapy. Tipifarnib was administered with food at a starting dose of 300 mg orally BID on Days 1 - 21 of 28-day treatment cycles.
  In the absence of unmanageable toxicity, treatment may have been continued as long as the investigator considered that the treatment was providing clinical benefit for up to 12 months since the subject's enrollment. Treatment may have continued beyond 12 months upon agreement by the investigator and sponsor if there was documented evidence of sustained clinical benefit.
- Cohort PTCL-NOS, CXCL12+: Subjects with PTCL-NOS CXCL12+ (not including subjects with PTCL-NOS) received tipifarnib as monotherapy. Tipifarnib was administered with food at a starting dose of 300 mg orally BID on Days 1 - 21 of 28-day treatment cycles.
  In the absence of unmanageable toxicity, treatment may have been continued as long as the investigator considered that the treatment was providing clinical benefit for up to 12 months since the subject's enrollment. Treatment may have continued beyond 12 months upon agreement by the investigator and sponsor if there was documented evidence of sustained clinical benefit.
- Cohort Other: Subjects with other indications (including ALCL-ALK negative and PTCL-subtype not specified per protocol) received tipifarnib as monotherapy. Tipifarnib was administered with food at a starting dose of 300 mg orally BID on Days 1 - 21 of 28-day treatment cycles.
  In the absence of unmanageable toxicity, treatment may have been continued as long as the investigator considered that the treatment was providing clinical benefit for up to 12 months since the subject's enrollment. Treatment may have continued beyond 12 months upon agreement by the investigator and sponsor if there was documented evidence of sustained clinical benefit.
Period: Overall Study
Arm/Group | Cohort AITL | Cohort PTCL-NOS | Cohort PTCL-NOS, CXCL12+ | Cohort Other
Started | 38 | 14 | 11 | 2
Completed | 2 | 0 | 0 | 0
Not Completed | 36 | 14 | 11 | 2
Not completed — Termination for Symptomatic Deterioration | 1 | 1 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 1 | 0
Not completed — Miscellaneous | 1 | 0 | 1 | 0
Not completed — Adverse Event | 9 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0
Not completed — Disease Progression | 22 | 12 | 5 | 2

BASELINE CHARACTERISTICS:
Population: The All Subjects as Treated (ASaT) Population consists of all enrolled subjects who received at least 1 dose of tipifarnib.
Groups:
- Cohort AITL: Subjects with AITL received tipifarnib as monotherapy. Tipifarnib was administered with food at a starting dose of 300 mg orally BID on Days 1 - 21 of 28-day treatment cycles.
  In the absence of unmanageable toxicity, treatment may have been continued as long as the investigator considered that the treatment was providing clinical benefit for up to 12 months since the subject's enrollment. Treatment may have continued beyond 12 months upon agreement by the investigator and sponsor if there was documented evidence of sustained clinical benefit.
- Total: Total of all reporting groups
Arm/Group | Cohort AITL | Cohort PTCL-NOS | Cohort PTCL-NOS, CXCL12+ | Cohort Other | Total
Number analyzed (Participants) | 38 | 14 | 11 | 2 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.50 (10.7) | 65.73 (13.7) | 65.74 (12.6) | 56.68 (12.0) | 65.32 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 2 | 5 | 1 | 24
  Male | 22 | 12 | 6 | 1 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 0 | 4
  Not Hispanic or Latino | 36 | 14 | 9 | 2 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 13 | 9 | 1 | 46
  Black or African American | 1 | 1 | 0 | 1 | 3
  Asian | 12 | 0 | 0 | 0 | 12
  Other | 2 | 0 | 2 | 0 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Score [Count of Participants; unit: Participants] — Performance Score:
  * 0: Fully active, able to carry on all predisease performance without restriction.
  * 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  * 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    Performance Score 0 | 18 | 3 | 5 | 0 | 26
    Performance Score 1 | 13 | 10 | 6 | 2 | 31
    Performance Score 2 | 7 | 1 | 0 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The ORR (complete response [CR] or partial response [PRs]) of tipifarnib was based on response assessments according to the Lugano Classification. Two-sided 95% confidence intervals (CIs) were based on either Wilson approximation (N > 4) or Clopper-Pearson method (N ≤ 4).
  CR: PET-CT-based response, score of 1-3 on five-point scale (5PS) for lymph nodes and extralymphatic sites, no evidence of fluorodeoxyglucose (FDG)-avid disease in marrow. CT-based response, target nodes and masses regress to 1.5 cm in longest transverse diameter, no extralymphatic sites of disease, normal bone marrow morphology.
  PR: PET-CT-based response, score of 4-5 on 5PS with reduced uptake compared to baseline for lymph nodes and extralymphatic sites, residual uptake reduced compared to baseline in the bone marrow. CT-based response, ≥ 50% decrease in sum of the product of perpendicular diameters of up to 6 target measurable nodes and extranodal sites, spleen regressed by > 50% in length beyond normal.
Time Frame: Up to approximately 3 years
Population: The Full Analysis Set (FAS) Population excluding subjects for the following reasons: no baseline data; failure to receive at least 1 dose of tipifarnib; no post-baseline endpoint data subsequent to at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort AITL | Cohort PTCL-NOS | Cohort PTCL-NOS, CXCL12+ | Cohort Other
Number analyzed (Participants) | 32 | 14 | 10 | 2
percentage of participants | 56.3 [39.3 to 71.8] | 7.1 [0.2 to 33.9] | 40.0 [12.2 to 73.8] | 0.0 [0.0 to 84.2]
Statistical Analysis 1: Comparison: Cohort AITL; Null hypothesis H0: PORR = 10% versus HA: PORR > 10% will be tested at a = 0.05 significance level using a two-sided binomial test. The choice of test statistics was driven by the method used for interval estimation; Test type: Other; p = 0.000, Wilson approximation
Statistical Analysis 2: Comparison: Cohort PTCL-NOS; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 1.000, Wilson approximation
Statistical Analysis 3: Comparison: Cohort PTCL-NOS, CXCL12+; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.026, Wilson approximation
Statistical Analysis 4: Comparison: Cohort Other; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 1.000, Clopper-Pearson method

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time (in months) from first dose (Cycle 1 Day 1) to either first observation of progressive disease (PD) or occurrence of death due to any cause within 126 days (approximately 2 time-intervals for tumor assessments) of either first administration of tipifarnib or the last tumor assessment. Observation of PD could have been by either documented radiographic progression (i.e., scan results) or documentation of symptomatic or clinical progression agreed upon and documented by investigators. In subjects without a progression date or with a death date more than 126 days after the first administration of study drugs or the last tumor assessment, the PFS time was censored on the date of last tumor assessment or date of first administration of study tipifarnib. The duration of the PFS was analyzed using the Kaplan-Meier (KM) method. 95% CIs were calculated using Hall-Wellner Method.
Time Frame: Up to approximately 3 years
Population: The FAS Population excluding subjects for the following reasons: no Baseline data; failure to receive at least 1 dose of tipifarnib; no post-baseline endpoint data subsequent to at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort AITL | Cohort PTCL-NOS | Cohort PTCL-NOS, CXCL12+ | Cohort Other
Number analyzed (Participants) | 32 | 14 | 10 | 2
months | 3.6 [1.9 to 8.3] | 2.1 [1.4 to 4.0] | 5.3 [1.8 to 11.1] | 1.4 [1.1 to 1.6]

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time (in months) from the start date of the objective response to the first date of either documented PD or death. No data imputations were conducted for missing data. In the event of a maintained response, the DOR was censored at the last evaluable non-PD assessment. The DOR was analyzed using the KM method. 95% CIs were calculated using Hall-Wellner Method.
Time Frame: Up to approximately 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort AITL | Cohort PTCL-NOS | Cohort PTCL-NOS, CXCL12+ | Cohort Other
Number analyzed (Participants) | 18 | 1 | 4 | 0
months | 7.8 [2.0 to 16.3] | 1.0 [NA to NA] — Lower 95% CI could not be estimated as there were too few participants with events that impacted the estimate of DOR function and there was no variation as per the pre-specified analysis in the SAP. | 2.8 [2.0 to NA] — Upper 95% CI was not reached as there were too few participants with events that impacted the estimate of DOR function. |

4. Secondary Outcome: Number of Subjects That Experienced One or More Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product, which did not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs that started on or after the first dose of study drug and within 30 days of the last administration of study drug or immediately before the initiation of any other anticancer therapy. The Investigator was required to grade the severity/intensity of each AE according to NCI-CTCAE version 4.03. If a severity/intensity of Grade 4 (life-threatening) or 5 (death) was applied to an AE, then the Investigator also reported the event as a serious AE.
Time Frame: Up to approximately 3 years
Population: The ASaT population consists of all enrolled subjects who received at least 1 dose of tipifarnib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort AITL | Cohort PTCL-NOS | Cohort PTCL-NOS, CXCL12+ | Cohort Other
Number analyzed (Participants) | 38 | 14 | 11 | 2
Participants
  TEAEs | 38 | 14 | 11 | 2
  Serious TEAEs | 21 | 8 | 8 | 1

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years
Arm/Group | Cohort AITL | Cohort PTCL-NOS | Cohort PTCL-NOS, CXCL12+ | Cohort Other
All-Cause Mortality (participants affected / at risk) | 13/38 | 8/14 | 4/11 | 1/2
Serious Adverse Events (participants affected / at risk) | 21/38 | 8/14 | 8/11 | 1/2
Other Adverse Events (participants affected / at risk) | 38/38 | 14/14 | 11/11 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort AITL (N=38) | Cohort PTCL-NOS (N=14) | Cohort PTCL-NOS, CXCL12+ (N=11) | Cohort Other (N=2)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Death (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Cytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort AITL (N=38) | Cohort PTCL-NOS (N=14) | Cohort PTCL-NOS, CXCL12+ (N=11) | Cohort Other (N=2)
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 8 | 2 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 3 | 3 | 3 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0
Chills (General disorders) | 4 | 1 | 2 | 1
Fatigue (General disorders) | 19 | 7 | 2 | 0
Gait disturbance (General disorders) | 2 | 1 | 0 | 0
Decreased activity (General disorders) | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 1 | 1 | 0
Malaise (General disorders) | 1 | 1 | 2 | 1
Oedema peripheral (General disorders) | 3 | 3 | 4 | 0
Pain (General disorders) | 2 | 0 | 1 | 1
Medical device pain (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 13 | 2 | 3 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 2 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 2 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 3 | 1 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 3 | 0 | 0
Blood creatinine increased (Investigations) | 5 | 5 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 1 | 0
Epstein-Barr virus test positive (Investigations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0 | 0
Human rhinovirus test positive (Investigations) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 4 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 0
Monocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 11 | 8 | 1 | 0
Platelet count decreased (Investigations) | 15 | 10 | 4 | 1
Urine output increased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 4 | 6 | 2 | 0
White blood cell count decreased (Investigations) | 4 | 3 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 16 | 10 | 6 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 4 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 8 | 2 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 5 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 5 | 5 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 14 | 8 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 5 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 12 | 9 | 4 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 5 | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 3 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urine abnormality (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 0 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 13 | 7 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 4 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 5 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 5 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 7 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 4 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 4 | 1 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 0 | 0
Streptoccocal urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There are agreements in place between clinical trial sites and the Sponsor (or its agents) that govern discussion or publication of trial results by the sites or their employees after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT02464228/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT02464228/SAP_001.pdf